CLINICAL TRIAL: NCT06009588
Title: Comparison of Self- and Balloon-expandable Valves in Patients With Ascending Aortic Dilation Undergoing Transcatheter Aortic Valve Replacement: The AAD-CHOICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-2024
Record Dates: First submitted 2023-08-12; First posted 2023-08-24 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Aortic Stenosis; Ascending Aortic Dilatation
Keywords: Transcatheter aortic valve replacement; Self-expandable valve; Balloon-expandable valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Self-expandable valve group vs. Balloon-expandable valve group
Who Masked: Participant, Investigator
Masking Description: Surgeons are aware of randomisation results, however, participants and research staff are all blinded to the randomisation schemes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-expandable valve group (Experimental): Patients using self-expandable valves
  Interventions: Device: self-expandable valves
- Balloon-expandable valve group (Experimental): Patients using balloon-expandable valves
  Interventions: Device: balloon-expandable valves

INTERVENTIONS:
Device: self-expandable valves — patients undergoing TAVR use self-expandable valves
  Arms: Self-expandable valve group
Device: balloon-expandable valves — patients undergoing TAVR use balloon-expandable valves
  Arms: Balloon-expandable valve group

SUMMARY:
This study aimed at comparing the performance of self-expandable valves versus balloon-expandable valves in patients with ascending aortic dilation undergoing transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
Ascending aortic (AA) dilation is a common feature in patients with aortic stenosis (AS), especially in those with bicuspid aortic valve (BAV). For patients undergoing surgical aortic valve replacement (SAVR), current guidelines recommend concomitant aortic repair or replacement if the diameter of AA exceeds 45mm to avoid aortic dissection or rupture.

Transcatheter aortic valve replacement (TAVR) has profoundly changed the clinical management of AS patients who cannot tolerate SAVR. For patients who are candidates for TAVR, simultaneous repair of a dilated AA can be technically difficult. The safety and feasibility of the procedure and the fate of AA after the procedure in these patients remain unclear. Moreover, there are limited data comparing the performance of self-expandable valves versus balloon-expandable valves in these patients. The aim of the present study is to evaluate the impact of type of transcatheter heart valves on intra-procedural device success and post-procedural AA progression in patients with dilated AA (≥45mm) undergoing TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis;
* Transfemoral access;
* Preoperative aortic CT suggesting maximum ascending aortic diameter ≥45mm and <55mm;
* Anticipated life expectancy >1 year;
* Age ≥ 65 years.

Exclusion Criteria:

* Dominant aortic regurgitation,;
* A history of SAVR or TAVR;
* A history of aortic surgery;
* Emergent TAVR.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | 30 days after TAVR procedure
  all-cause mortality within 30 days after TAVR procedure
30-day adverse aortic events | 30 days after TAVR procedure
  aortic death, aortic dissection, or aortic rupture
The rate of device success | 30 days
  Device success is defined as following:
  1. Technical success (Freedom from mortality; Successful access, delivery of the device, and retrieval of the delivery system; Correct positioning of a single prosthetic heart valve into the proper anatomical location; Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication)
  2. Freedom from mortality
  3. Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  4. Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index $0.25, and less than moderate aortic regurgitation)

SECONDARY OUTCOMES:
1-year all-cause mortality | 1 year after TAVR procedure
  all-cause mortality
1-year cardiovascular mortality | 1 year after TAVR procedure
  Related to heart failure, cardiogenic shock, bioprosthetic valve dysfunction, myocardial infarction, stroke, thromboembolism, bleeding, tamponade, vascular complication, arrhythmia or conduction system disturbances, cardiovascular infection (e.g. mediastinitis, endocarditis), or other clear cardiovascular cause
1-year adverse aortic events | 1 year after TAVR procedure
  aortic death, aortic dissection, or aortic rupture
Ascending aortic diameter expansion rate ≥3mm/year | 1 year after TAVR procedure
  Expansion rate was calculated as the change of ascending aortic diameters (before the procedure and at the latest follow-up) divided by the follow-up period.
Hospitalization (or re-hospitalization) | 1 year after TAVR procedure
  Any admission after the index hospitalization or study enrolment to an inpatient unit or hospital ward for ≥24 h, including an emergency department stay.
  Hospitalizations planned for pre-existing conditions are excluded unless there is worsening of the baseline condition. Visits to urgent care centres or emergency departments <24 h may also be included if substantive intensification of therapy changes (e.g. heart failure episodes) are enacted (e.g. intravenous diuretics, significant increases in drug therapy dosages or addition of new pharmacotherapy agents)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD, Principal Investigator — Department of Structural Heart Disease, National Center for Cardiovascular Disease, China & Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- National Center for Cardiovascular Disease, China & Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VARC-3 WRITING COMMITTEE:; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: Updated Endpoint Definitions for Aortic Valve Clinical Research. J Am Coll Cardiol. 2021 Jun 1;77(21):2717-2746. doi: 10.1016/j.jacc.2021.02.038. Epub 2021 Apr 19. PMID 33888385
- [Derived] An K, Zhang F, Ouyang W, Li S, Pan X. Protocol for a randomized controlled trial for comparison of self- and balloon-expandable valves in patients with Ascending Aortic Dilation Undergoing Transcatheter Aortic Valve Replacement (AAD-CHOICE). Trials. 2025 Nov 28;27(1):1. doi: 10.1186/s13063-025-09233-7. PMID 41316413